CLINICAL TRIAL: NCT01412684
Title: Pilot Study of Distal Pancreatectomy With Partial Splenectomy for Pancreatic Tumors Arising in the Body and Tail of the Pancreas
Brief Title: Distal Pancreatectomy With Partial Splenectomy for Pancreatic Tumors
Status: Withdrawn | Type: Observational
Why Stopped: Never activated
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: MU1196577
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-05

CONDITIONS: Tumor of Exocrine Pancreas
MeSH Terms: interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Distal pancreatectomy with partial splenectomy — Distal pancreatectomy with partial splenectomy
  Other Names: pancreatectomy

SUMMARY:
Most resectable tumors arising in the body or tail of the pancreas are malignancies or premalignancies which are surgically treated with distal pancreatectomy in combination with splenectomy. Retrieval of the lymph node tissue which lies along the splenic vessels is necessary to complete an oncologically sound operation. Two techniques for spleen preserving distal pancreatectomy have been described, but only a small number of lesions are amenable to spleen preserving pancreas surgery because these operation compromise oncologic principles. Removal of a normal spleen usually does not cause immediate consequences but can make patients vulnerable to life threatening infections. Asplenic patients must be vigilant for these infections and antibiotic prophylaxis is recommended anytime a fever occurs. Splenectomy results in measurable changes in the cellular components of the blood. If thrombocytosis occurs as a result of splenectomy, it requires life-long antiplatelet treatment.

Some childhood hematologic disorders such as hereditary spherocytosis are successfully treated with partial splenectomy. The post-surgical remnant spleen has been shown to be viable and functional. Both hematologic and immunologic function of the spleen seems to be preserved in most patients. Partial splenectomy has also been successful ly employed to treat benign and malignant lesions of the spleen. Unfortunately these indications for surgery are rare and so the experience with partial splenectomy is small.

To date, distal pancreatectomy with partial splenectomy has not been described in the medical literature. The investigators have devised a surgical procedure combining distal pancreatectomy with partial splenectomy, in principal allowing preservation of splenic function without compromise of oncologic principles. This procedure is possible now because of new technology which allows for near bloodless transection of solid organs. These instruments are routinely used in liver, kidney and pancreas surgery. There are scattered reports of successful use of these instruments in splenic transection, but there is no large experience to date.

The study intends to answer the question, is the proposed procedure, distal pancreatectomy and partial splenectomy, a viable alternative to the current standard of care, distal pancreatectomy with total splenectomy, for patients who will undergo surgical treatment of pancreas lesions arising in the body or tail of the pancreas?

DETAILED DESCRIPTION:
Resectable tumors arising in the body or tail of the pancreas are malignancies or premalignancies which are surgically treated with distal pancreatectomy in combination with splenectomy. Retrieval of the lymph node tissue which lies along the splenic vessels is necessary to complete an oncologically sound operation. Two techniques for spleen preserving distal pancreatectomy have been described, but only a small number of lesions are amenable to spleen preserving pancreas surgery because these operation compromise oncologic principles. Removal of a normal spleen usually does not cause immediate consequences but can make patients vulnerable to life threatening infections. Asplenic patients must be vigilant for these infections and antibiotic prophylaxis is recommended anytime a fever occurs. Splenectomy results in measurable changes in the cellular components of the blood. If thrombocytosis occurs as a result of splenectomy, it requires life-long antiplatelet treatment.

Some childhood hematologic disorders such as hereditary spherocytosis are successfully treated with partial splenectomy. The post-surgical remnant spleen has been shown to be viable and functional. Both hematologic and immunologic function of the spleen seems to be preserved in most patients. Partial splenectomy has also been successful ly employed to treat benign and malignant lesions of the spleen. Unfortunately these indications for surgery are rare and so the experience with partial splenectomy is small.

To date, distal pancreatectomy with partial splenectomy has not been described in the medical literature. We have devised a surgical procedure combining distal pancreatectomy with partial splenectomy, in principal allowing preservation of splenic function without compromise of oncologic principles. This procedure is possible now because of new technology which allows for near bloodless transection of solid organs. These instruments are routinely used in liver, kidney and pancreas surgery. There are scattered reports of successful use of these instruments in splenic transection, but there is no large experience to date.

The study intends to answer the question, is the proposed procedure, distal pancreatectomy and partial splenectomy, a viable alternative to the current standard of care, distal pancreatectomy with total splenectomy, for patients who will undergo surgical treatment of pancreas lesions arising in the body or tail of the pancreas?

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid or cystic neoplasms of the pancreas who are being considered for distal pancreatectomy/splenectomy to be performed in either an open, laparoscopic, of da Vinci assisted fashion.
* No evidence of metastatic disease
* No evidence of local invasion into surrounding organs
* ECOG performance status <3
* Age 18 years or greater
* Participants will provide written informed consent to be part of the study

Exclusion Criteria:

* Age less than 18 years old
* Women who are pregnant
* Known hereditary bleeding disorder with history of post-operative hemorrhage
* Patients maintained on chronic anticoagulation (eg Coumadin therapy)
* Known hematogenous disorder
* Previous gastric fundoplication procedure or any procedure which interrupts the short gastric blood supply to the spleen
* Known primary or secondary malignancy of the spleen
* Pancreatic tumors which invade surrounding structures
* Prisoners
* Patients with impaired decision-making skills

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: surgical oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Splenic function | 30 days post-operatively

SECONDARY OUTCOMES:
Lymph node retrieval | within 30 days post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nicholl, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States